CLINICAL TRIAL: NCT05904535
Title: Novel Diagnostic Methods to Identify External Ventricular Drain Associated Infections
Acronym: EVD Infect II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Region Stockholm (Other Government); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, David Nelson, MD , PhD, MD, PhD, Karolinska University Hospital
Other Study IDs: K 2022-7809
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Ventricular Drain Related Infection; Nosocomial Infection; Infection, Bacterial; Ventriculitis, Infectious
MeSH Terms: conditions — Cross Infection; Bacterial Infections; Cerebral Ventriculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid from external ventricular drains.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Cerebrospinal fluid will be collected from all study subjects and analyzed with sequencing techniques, Optotracing, and REDOX. All methods will compared with CSF bacterial cultures which is the current golden standard.
  Interventions: Other: Cerbrospinal fluid sampling.

INTERVENTIONS:
Other: Cerbrospinal fluid sampling. — Routine sampling of cerebrospinal fluid from the proximal external ventricular drain port.

SUMMARY:
External ventricular drain infections are difficult to identify with current diagnostic methods. Initiation of antibiotic treatment is usually supported by indirect methods of bacterial infection, such as clinical signs or cerebrospinal fluid cell counts (CSF). As such, excessive treatment with antibiotics is common in these patients due to suspected infection while the incidence of true culture confirmed infections are less common. This study will evaluate three novel diagnostic methods for rapid direct bacterial detection in CSF, in order to assess if these can be used to guide antibiotic treatment in neurocritically ill patients, compared to CSF bacterial cultures.

DETAILED DESCRIPTION:
In the literature, the reported incidence ranges between 1-35% of inserted drains. This disparity results from the lack of an international consensus on a definition for EVDIs and the use of various diagnostic criteria across studies. In a neurointensive care setting, clinical symptoms are often difficult to evaluate due to underlying illness. Cerebrospinal fluid (CSF) bacterial culture is the current golden standard of EVDI diagnostics. However, CSF bacterial cultures often take several days to finalize and prior use of antibiotics may further prolong culture incubation time or cause false negative cultures. It is seldom possible to delay treatment until the bacterial cultures have finalized. Additionally, due to the etiology of these infections, contamination and true positives can be difficult to distinguish based on the cultured bacteria alone. Thus, early identification of EVDIs are based on indirect signs of bacterial infection, namely CSF analysis of glucose, lactate, protein, leukocytes, and erythrocytes. In the neurocritically ill, CSF parameters are frequently confounded by intraventricular hemorrhage (IVH). Leukocytes and erythrocytes in particular may vary greatly depending on the IVH volume.

To adjust for IVH, the ratio of leukocytes and erythrocytes (LE ratio) in CSF is commonly used and is one of the main metrics in identifying EVDIs. The LE ratio is based on the assumption that erythrocytes and leukocytes are homogeneously distributed in the CSF. This assumption has previously not been questioned. However, it is clear from computed tomography (CT) scans that blood sediments in the ventricles, suggesting that a homogeneous distribution is unlikely. The LE ratio fails to account for the fact that the blood causes an aseptic inflammation in itself, resulting in immigration of leukocytes. Additionally, leukocytes, in particular granulocytes, may exhibit upwards floatation, or antisedimentation, a property shown to be exacerbated in critically ill patients. Thus, leukocytes may sediment at a slower rate than erythrocytes which may further skew the intraventricular CSF/blood distribution towards heterogeneity.

Due to the specific pathogens, patient characteristics, and confounding factors, early identification of EVDIs have proven difficult and no CSF parameter, by itself or in aggregate, have yet been shown to reliably predict or identify EVDIs. As such, algorithms based on routinely analyzed CSF parameters and clinical symptoms are ambiguous and diagnosis is often based on "expert-opinion". This results in an excessive use of broad spectrum antibiotics and a large variation in clinical practice, with up to 10-20 patients being treated for every true infection. Additionally, the main metric in EVDI diagnostics, the LE ratio, is based on the uncertain assumption that cells are homogeneously distributed in the CSF. If, and how, this affects routinely analyzed CSF parameters has yet to be studied. With the questionable precision of current indirect methods to identify EVDIs in mind, there is a need for more rapid and accurate tools for direct microbiological detection and identification in the diagnostics of EVDI.

The use of emerging bacterial DNA sequencing techniques in infectious diseases medicine increasing. Unfortunately, these techniques for CSF with primers covering the specific bacteria found in EVDIs have not yet been verified. Moreover, due to the lack of established around the clock work flows surrounding these methods, results from these techniques are not yet readily available within the time-frame needed to decide whether to instigate treatment. However, regular PCR methods have been shown to identify bacteria in a large portion of clinically suspected severe sepsis patients exhibiting negative blood cultures. Interestingly, this group had the highest mortality suggesting that the positive bacterial findings were not just due to the use of an oversensitive technique. Bacterial DNA sequencing techniques may have the potential to exhibit a higher sensitivity compared to conventional bacterial cultures within a smaller time frame.

16s ribosomal ribonucleic acid (16s rRNA) is a component of the prokaryotic ribosomal 30s subunit and is present in all prokaryotic lifeforms. The use of 16s rRNA sequencing have been shown to reliably identify bacteria in normally sterile body fluids, such as CSF, compared to bacterial cultures. 16s rRNA also have the advantage of being able to identify non viable bacteria, thus potentially exhibiting a greater sensitivity in patients who have been subjected to antibiotic treatment prior to sampling, making it a promising target for bacterial DNA sequencing. However, 16s rRNA sequencing have not been studied extensively for EVDIs.

Optotracing is a novel method for identification of bacteria and bacterial biofilms. The method is based on luminescent conjugated oligothiophenes (LCOs), a polymer which exhibit optoelectric properties. Interaction between LCOs and biofilm products or bacteria directly lead to target specific fluorescent emission which allows for optical detection. The method have recently been found to reliably identify biofilm producing uropathogenic E. Coli in patients with urinary tract infection. Furthermore, the method was able to differentiate between healthy and infected urine regardless of the detection of biofilm products. Optoelectric polymers are versatile molecules enabling easy modification which may allow for tailored target specific interaction, potentially allowing optotracing to be used as a method for specific rapid bacterial identification in EVDI diagnostics.

In addition to optotracing, electrochemical sensing of bacterial metabolic activity (REDOX) have recently been investigated as a new method of bacterial detection. REDOX exploits the reducing capabilities of bacteria. This property have enabled the creation of a rapid, highly sensitive test array using polymers with semiconductive properties acting as an electron acceptor. This method allows for the measurement of the metabolic activity of bacteria in real-time by measuring the current induced by direct transfer of electrons from the bacteria to the polymer surface or indirectly, by release of redox active compounds. The use of conducting and optoeletric polymers to detect bacteria represents an exiting new field of research with promising clinical applications that may enable direct, precise, and rapid microbiological diagnostics and allow for real-time surveillance of bacterial growth.

The overall aim of this project is to study novel methods of direct bacterial detection in EVDI diagnostics to evaluate if these methods can be used to guide treatment in order to reduce excessive treatment with broad-spectrum antibiotics in neurocritically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Treated with an external ventricular drain.
2. Admitted to the neurocritical and critical care unit at Karolinska University Hospital in Solna, Sweden.

Exclusion Criteria:

1. Does not fulfill age requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a minimum age of 18, who are admitted to the ICU and treated with an external ventricular drain. All patients will be included regardless of underlying admission diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Specificity | 2022-2025
  Each methods specificity will be prospectively evaluated.

SECONDARY OUTCOMES:
Sensitivity | 2022-2025
  Each methods sensitivity will be prospectively evaluated. Due to the low incidence of true infections the sensitivity will mainly be evaluated using spiked CSF samples.

CONTACTS AND LOCATIONS:
Overall Officials: David W Nelson, MD, PhD, Principal Investigator — Karolinska University Hospial, Karolinska Institutet
Locations (1):
- Perioperative Medicine and Intensive Care, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to 10 years after manuscript publication.
Access Criteria: Shared upon reasonable request to study officials.